CLINICAL TRIAL: NCT03258983
Title: Alpha-linolenic Acid and the Risk of Atherosclerotic Cardiovascular Disease
Brief Title: Alpha-linolenic Acid and the Risk of ASCVD
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Christian Sørensen Bork, Dr. Christian Sørensen Bork, Aalborg University Hospital
Other Study IDs: 17-R115-A7415-22060 - 2016-229
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Acute Myocardial Infarction; Ischemic Stroke; Peripheral Artery Disease
Keywords: Alpha-linolenic acid; Dietary intake; Adipose tissue; Nutritional epidemiology
MeSH Terms: conditions — Ischemic Stroke; Peripheral Arterial Disease | interventions — alpha-Linolenic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subcutaneous adipose tissue, serum, plasma, ''buffycoat'', erytrocytes and urine is stored in nitrogen vapour at the biobank of the Diet, Cancer and Health cohort study. Also, whole blood in filter paper and toenail clippings has been stored within the biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Diet, Cancer and Health cohort
  Interventions: Other: Alpha-linolenic acid

INTERVENTIONS:
Other: Alpha-linolenic acid — Exposure to dietary intake of alpha-linolenic acid (ALA) will be assessed using a detailed food frequency questionaire filled in by participants included in the Diet, Cancer and Health cohort at baseline. Exposure to adipose tissue content of ALA will be determined by gas chromatography in all incident cases and in subcohort of 3500 participants randomly drawn from the total cohort.
  Other Names: ALA (18:3-n3)

SUMMARY:
Background: The plant-derived omega-3 fatty acid alpha-linolenic acid (ALA, 18:3-n-3) may reduce the risk of atherosclerotic cardiovascular disease, including incident myocardial infarction, ischemic stroke and peripheral artery disease. However, the results of previous studies have been inconsistent.

Objectives: To investigate the associations between dietary intake of ALA, adipose tissue content of ALA, and the risk of the major atherosclerotic cardiovascular diseases incident myocardial infarction, ischemic stroke and subtypes, and peripheral artery disease.

Methods: This project will be based on data from the Danish cohort study Diet, Cancer and Health which consisted of 57,053 men and women at recruitment between 1993 and 1997. Dietary intake of ALA will be assessed using a validated semiquantitative food-frequency questionnaire and adipose tissue content will be determined with the use of gas chromatography analyses of adipose tissue biopsies collected at baseline. Also, detailed information on lifestyle factors, medical history and anthropometri was collected at baseline.

Incident cases have been identified through national registries and the diagnoses have previously been validated.

Analyses of dietary intake of ALA will be analysed using a traditional cohort design, whereas analyses on adipose tissue content of ALA will be analysed based on a case-cohort design. Hazard ratioes with 95% confidence intervals will be used to describe the associations between the exposure variables and the outcome variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Born in Denmark
* Age between 50 and 64 years
* Living in the areas of Copenhagen and Aarhus

Exclusion Criteria:

* Previous cancer

Ages: 50 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The Diet, Cancer and Health cohort was established over a period of 3.5 years between 1993 and 1997 by inviting 160,725 men and women to participate. All eligible participants were native Danish citizens without a previous diagnosis of cancer, aged 50-64 years, and living in the areas of Copenhagen and Aarhus. A total of 57053 accepted to participate in the Diet, Cancer and Health cohort study.
  A subcohort of 3500 participants were drawn randomly from the cohort at baseline.
Sampling Method: Probability Sample
Enrollment: 57053 (Actual)
Dates: Start 1993-11-24 (Actual); Primary Completion 2013-07-10 (Actual); Study Completion 2013-07-10 (Actual)

PRIMARY OUTCOMES:
Incident acute myocardial infarction | From baseline until July 2013
Incident ischemic stroke including total and subtypes of ischemic stroke | From baseline until November 2009
Incident peripheral artery disease | From baseline until December 2009

SECONDARY OUTCOMES:
Incident fatal myocardial infarction | From baseline until July 2013

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Bork, MD, Principal Investigator — Department of Cardiology, Aalborg University Hospital, Denmark

REFERENCES:
- [Background] Tjonneland A, Olsen A, Boll K, Stripp C, Christensen J, Engholm G, Overvad K. Study design, exposure variables, and socioeconomic determinants of participation in Diet, Cancer and Health: a population-based prospective cohort study of 57,053 men and women in Denmark. Scand J Public Health. 2007;35(4):432-41. doi: 10.1080/14034940601047986. PMID 17786808
- [Derived] Bork CS, Veno SK, Lundbye-Christensen S, Jakobsen MU, Tjonneland A, Schmidt EB, Overvad K. Dietary Intake of alpha-Linolenic Acid Is Not Appreciably Associated with Risk of Ischemic Stroke among Middle-Aged Danish Men and Women. J Nutr. 2018 Jun 1;148(6):952-958. doi: 10.1093/jn/nxy056. PMID 29767732